CLINICAL TRIAL: NCT06164509
Title: Healing Potentiality of Different Doses of Trypsin and Alpha Chemo Trypsin in Mandibular Molars With Chronic Apical Abscess
Brief Title: Healing Potentiality of Trypsin and Alpha Chemo Trypsin in Mandibular Molars With Chronic Apical Abscess
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AinShamsUNII
Record Dates: First submitted 2023-11-21; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-11

CONDITIONS: Mandibular Abscess
MeSH Terms: interventions — Tablets; Extravehicular Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Alphintern (Active Comparator): Group A will receive (Alphintern® tablet, Amoun, Egypt),
  Interventions: Drug: Alphintern® , tablet, Amoun, Egypt
- Alzyme Max (Active Comparator): Group B will receive (Limitless Allzyme Max®, tablet, Eva, Egypt)
  Interventions: Drug: Alphintern® , tablet, Amoun, Egypt
- Placebo (No Intervention): Group C will not receive medication

INTERVENTIONS:
Drug: Alphintern® , tablet, Amoun, Egypt — Medications will be taken three times daily for 7 days postoperative, after that all cases will be reexamined regarding healing rate, adverse effect and failure rate of medical treatment.
  Other Names: Limitless Allzyme Max®, tablet, Eva, Egypt
  Arms: Alphintern; Alzyme Max

SUMMARY:
assessment of healing potentiality of peri apical lesions using different doses of trypsin and alpha chemo trypsin in mandibular molars with chronic apical abscess

DETAILED DESCRIPTION:
Owing to anti-inflammatory, anti-oedematous, fibrinolytic, anti-infective, and analgesic effects, trypsin:

chymotrypsin oral combination has emerged as a promising treatment of mandibular molars with chronic apical abscess. Trypsin chymotrypsin combination always showed a significant reduction in swelling and pain postoperatively.

Study procedures:

1. According to inclusion and exclusion criteria; patients will be subjected to complete history taking, general and local "dental" examinations.
2. Important dental symptoms will be assessed include bleeding, pain, malocclusion, new growths, numbness or paresthesias, and chewing problems.
3. General information will be reported including use of alcohol or tobacco and systemic symptoms, such as fever and weight loss.
4. A thorough inspection with good illumination, a tongue blade, gloves, and a gauze pad will be performed.
5. Complete or partial dentures will be removed so that underlying soft tissues can be seen.
6. A head-mounted light will be used. However, because the light cannot be precisely aligned on the axis of vision, it is difficult to avoid shadowing in narrow areas.
7. Better illumination results will be performed with a head-mounted convex mirror.
8. The temporomandibular joint (TMJ) will be assessed by looking for jaw deviation on opening and by palpating the head of the condyle anterior to the external auditory meatus.
9. Examiner then place his little fingers into the external ear canals with the pads of the fingertips lightly pushing anteriorly while patients repeatedly open widely and then close.
10. Preoperative preapical X-ray and CBCT will be done.
11. Cases will be randomly divided into 3 groups; Group A will receive (Alphintern®, tablet, Amoun, Egypt), Group B will receive (Limitless Allzyme Max®, tablet, Eva, Egypt) Group C will not receive medication
12. Medications will be taken three times daily for 7 days postoperative, after that all cases will be reexamined regarding healing rate, adverse effect and failure rate of medical treatment.
13. Randomization, allocation and concealment: It will be done using computer generated randomization sheet. Sealed opaque packages will be given to a third person (nurse) who will assign the packages to study groups. Each patient will be invited to pull out a package. According to the number inside package, cases will be allocated to either group A, B or C according to a computer- generated random list.
14. Postoperative preapical X-ray will be done at the end of the root canal treatment.
15. Patient will be recalled after three months for preapical X-ray assessment.
16. After six months patient will be recalled for preapical X-ray and CBCT to be done.

ELIGIBILITY:
Inclusion Criteria:

1. Age: any age group.
2. Both genders.
3. Cases with mandibular molars with chronic apical abscess

Exclusion Criteria:

1. Patients with significant comorbidities like uncontrolled diabetes mellitus, hypertension, hepatic or renal disorders.
2. Immunocompromised patients.
3. Patient with allergy from study medications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Lesion size and bone Formation will be measured by cone-beam computed tomography | 6 months
  cone-beam computed tomography will be done Before Drug is given and after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Nasir City, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouillaguet S, Manoil D, Girard M, Louis J, Gaia N, Leo S, Schrenzel J, Lazarevic V. Root Microbiota in Primary and Secondary Apical Periodontitis. Front Microbiol. 2018 Oct 9;9:2374. doi: 10.3389/fmicb.2018.02374. eCollection 2018. PMID 30356779
- [Background] Oberoi SS, Dhingra C, Sharma G, Sardana D. Antibiotics in dental practice: how justified are we. Int Dent J. 2015 Feb;65(1):4-10. doi: 10.1111/idj.12146. Epub 2014 Dec 16. PMID 25510967